CLINICAL TRIAL: NCT05143645
Title: Evaluation of a New Clinical Protocol for Dose Selection of Vancomycin for Continuous Infusion in ICU Patients.
Brief Title: A New Protocol for Continuous Vancomycin Infusion Dosing.
Acronym: CVIP
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Petersson, Senior ICU Consultant, Karolinska University Hospital
Other Study IDs: K 2019-9605
Record Dates: First submitted 2019-11-03; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Sepsis; Vancomycin Treatment
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Plasma vancoymcin measurements

SUMMARY:
This observational study prospectively collect data on chosen dosing, renal function, measured plasma concentrations and adherence to the recommended clinical protocl for ICU patients treated with continuous vancomycin infusion.

ELIGIBILITY:
Inclusion Criteria:

- Start of continuous vancomycin infusion during the course of intensive care and at least one measurement of plasma concentration.

Exclusion Criteria:

* Vancomycin treatment within 96 h before admission to the unit.
* Vancomycin treatment started with intermittent bolus infusions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ICU patients.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Time (days) from start of treatment to first measurement of a plasma vancomycin concentration between 20 and 25 mg/mL | Until the end of treatment or discharge from unit
  The title is a full description.
Relationship between time to intended concentration (15-20 mg/L) and adherence to the dosing protocol (% complete adherence). | Until the end of treatment or discharge from unit
  For each patient the actually administired dose of vancomycin will be compared to the recommendation in the dosing protocol. The time to the intended concentration will be compared between patients with 100% adherence to the recommendations and for patients with dosing not following the recommendations.

SECONDARY OUTCOMES:
Percentage of the total treatment duration with the intended plasma concentration 15-20 mg/L. | Until the end of treatment or discharge from unit
  The title is a full description.
Relationship between Percentage of the total treatment duration with the intended plasma concentration (15-20 mg/L) and adherence to the dosing protocol. | Until the end of treatment or discharge from unit
  The title in combination with the description of outcome 2 is a sufficient description.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided